CLINICAL TRIAL: NCT01042938
Title: Curcumin for the Prevention of Radiation-induced Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Julie Ryan, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URCC1106; 5KL2RR024136-03 (NIH); 05-238-80 (Other Grant/Funding Number: Dermatology Foundation)
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: Radiation dermatitis in breast cancer patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Curcumin; Diarylheptanoids; calcium phosphate, dibasic, dihydrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin C3 Complex (Active Comparator): Patients take 2.0 grams curcumin (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (~4-7 weeks).
  Interventions: Drug: Curcumin C3 Complex
- Placebo (Placebo Comparator): Patients take 2.0 grams placebo (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (~4-7 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin C3 Complex — Patients take 2.0 grams curcumin (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (~4-7 weeks)
  Other Names: Curcumin; curcuminoids
  Arms: Curcumin C3 Complex
Drug: Placebo — Patients take 2.0 grams placebo (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (~4-7 weeks)
  Other Names: dicalcium phosphate with yellow food grade dye
  Arms: Placebo

SUMMARY:
Ionizing radiation is a toxic agent and widely accepted form of treatment for various types of cancer. Despite advances in medical technology, radiation therapy still causes severe early and late skin effects. Radiation-induced dermatitis occurs in approximately 80% of patients. Important consequences of radiation-induced dermatitis include impairment of the quality of a patient's life due to pain and premature interruption of radiation treatment, which in turn, may be impair good local control of disease. The biological pathways responsible for acute radiation-induced dermatitis remain unclear. Currently, there is no standard treatment for the prevention of radiation-induced dermatitis with demonstrated effectiveness. The aim of this randomized, double-blind, placebo-controlled pilot study is to assess the effectiveness of curcumin for the prevention of acute radiation-induced dermatitis during postoperative radiotherapy for breast cancer. We hypothesize that curcumin, a natural phenolic compound found in both turmeric and curry powders, can prevent or alleviate radiation-induced skin reactions in breast cancer patients receiving radiotherapy.

DETAILED DESCRIPTION:
Specifically, this clinical pilot study will develop data necessary to calculate a sample size for a larger study to be conducted through the National Cancer Institute (NCI) Community Clinical Oncology Program (CCOP) mechanism. Specifically, this pilot project will investigate: 1) if curcumin can prevent or alleviate radiation-induced skin reactions in cancer patients receiving radiotherapy and 2) if skin pigmentation, as well as pain and psychophysiological factors, can predict the severity of radiation-induced dermatitis. Potential future research studies may be conducted to identify the biological mechanisms involved in radiation-induced dermatitis and the radioprotective function of curcumin.

ELIGIBILITY:
Inclusion Criteria:

* Female with a diagnosis of, non-inflammatory breast adenocarcinoma and be referred for post-operative radiotherapy without concurrent chemotherapy.
* Participants must be at least 21 years of age.
* Participants must not be pregnant.
* Participants can be from any racial or ethnic origin.
* Breast adenocarcinoma could have been treated by either lumpectomy or mastectomy with or without adjuvant or neoadjuvant chemotherapy or hormonal treatment.
* Participants with in situ breast cancer are eligible.
* Participants who are prescribed concurrent hormone treatment with radiation treatment are eligible.
* Participants must be scheduled to receive five sessions of radiation therapy per week (1 session per day) for at least four weeks using standard (1.8-2.0 Gy per session)or Canadian (2.2-2.5 Gy per session)irradiation fractionation.
* A time period of three weeks must elapse after chemotherapy and surgery before beginning the study.
* The total dose prescribed to the whole breast should be 50 Gy or greater.
* Participants must be able to understand English and able to complete assessment forms (all assessment forms are in English).
* Participants must be able to swallow medication.
* Topical skin agents, e.g., Aquaphor, Cetaphil, or other emollients, are allowed either PRN or prophylactically.
* Participant must give informed consent.

Exclusion Criteria:

* Patients with bilateral breast cancer are not eligible.
* Patients who have had previous radiation therapy to the breast or chest are not eligible.
* Patients who are prescribed chemotherapy concurrently with radiation treatment are not eligible.
* Patients who will be receiving treatment with Herceptin (trastuzumab), anti-coagulants, or anti-human epidermal growth factor receptor (EGFR) drugs, e.g. Iressa (gefitinib), Erbitux (cetuximab, C225), concurrently with their radiation therapy are not eligible.
* Patients cannot have had breast reconstructions, implants, and/or expanders.
* Patients with known radiosensitivity syndromes (e.g., Ataxia-telangiectasia) are not eligible.
* Patients with collagen vascular disease, vasculitis, unhealed surgical sites, or breast infections are not eligible.
* Patients whose baseline blood tests meet the following criteria are not eligible: greater than or equal to Grade 2 change Hemoglobin (i.e., 25% decrease from baseline); greater than or equal to Grade 1 change in Platelets (i.e., less than 75,000/mm3); greater than or equal to Grade 2 change in PT and PTT(i.e., 1.5-2x upper level normal (ULN)); greater than or equal to Grade 1 change in AST, ALT (i.e., greater than 2.5x ULN); greater than or equal to Grade 1 change in Bilirubin (i.e., greater than 1.5x ULN); greater than or equal to Grade 1 change in Creatinine (i.e., greater than 2x ULN).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Ryan, PhD, MPH, Principal Investigator — University of Rochester Medical Center & Wilmot Cancer Center; Julie L Ryan, PhD, MPH, Study Chair — University of Rochester Medical Center & Wilmot Cancer Center; Alice P Pentland, MD, Study Chair — University of Rochester Medical Center & Wilmot Cancer Center; Marilyn Ling, MD, Study Chair — University of Rochester Medical Center & Wilmot Cancer Center
Locations (1):
- University of Rochester Medical Center & Wilmot Cancer Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this trial began January 18, 2008 and ended on January 27, 2010. All patients were recruited and treated at the University of Rochester Cancer Center. Of the 213 breast cancer patients prescribed radiation therapy during this timeframe, 67 patients were approached for particiaption in the trial.
Period: Overall Study
Arm/Group | Curcumin C3 Complex | Placebo
Started | 17 (1 withdrew before radiation; 1 ineligible due to other clinical trial; 1 non-compliance.) | 18 (1 withdrew before radiation; 1 non-compliance.)
Completed | 14 | 16
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Ineligible: RTOG study conflict | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin C3 Complex | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 2 | 5 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 50.4 (9.51) | 53.7 (7.55) | 51.8 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Severity of Dermatitis in Radiation Treatment Site in Breast Cancer Patients
Description: The severity of radiation dermatitis was measured using the Radiation Dermatitis Severity (RDS)Scale which ranges from 0.0 to 4.0 with increments of 0.5. The RDS scale is a revised form of the NIH Common Toxicity Criteria to account for color and subtle texture changes in the skin. The worst dermatitis (i.e., highest RDS score) at the end of treatment was used for the primary analysis of severity of radiation dermatitis in each treatment group. Additionally, we performed repeated measure analyses to examine the severity of dermatitis over time in each arm.
Time Frame: 4-7 weeks (prescribed course of radiation)
Population: We used all 30 participants that fully completed the trial in all of our analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Curcumin C3 Complex: Patients take 2.0 grams curcumin (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (RT) (~4-7 weeks).
- Placebo: Patients take 2.0 grams placebo (four 500mg capsules) three times daily by mouth for prescribed course of radiation treatment (RT)(~4-7 weeks).
Arm/Group | Curcumin C3 Complex | Placebo
Number analyzed (Participants) | 14 | 16
units on a scale | 2.6 (0.994) [2.06 to 3.15] | 3.4 (0.554) [3.11 to 3.70]
Statistical Analysis 1: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: The mean RDS for curcumin group is significantly different (i.e., lower) than mean RDS of placebo group at end of radiation treatment; Test type: Superiority or Other; p = 0.0077, Standard pooled variances t-test; Mean Difference (Final Values) = -0.7991, 95% CI 2-sided [-1.3693 to -0.2289], Standard Deviation 0.7606

2. Secondary Outcome: Moist Desquamation at Radiation Treatment Site
Description: The presence of moist desquamation at the end of radiation treatment was examined between curcumin and placebo treatment groups. We compared the number of participants (or percentage) with moist desquamation between each treatment group.
Time Frame: 4-7 weeks (prescribed course of radiation)
Population: All 30 participants who completed the trial were used in all analyses.
Measure: Number; unit: participants
Arm/Group | Curcumin C3 Complex | Placebo
Number analyzed (Participants) | 14 | 16
participants | 4 | 14
Statistical Analysis 1: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: The presence of moist desquamation significantly differed between the curcumin group and the placebo group; Test type: Superiority or Other; p = 0.0022, Fisher Exact

3. Secondary Outcome: Redness at Radiation Treatment Site
Description: Redness at radiation treatment site was measured using a CR-400 Colorimeter (Konica Minolta). The colorimeter uses the L*a*b* color scale. We used a* values (redness) which range from 0.0 to 20.0. The lower the number value, the lower amount of redness. Therefore, high number values represent large amounts of redness.
Time Frame: 4-7 weeks (prescribed course of radiation)
Population: The 30 participants that fullt completed the trial were used in these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale (0.0 to 20.0)
Arm/Group | Curcumin C3 Complex | Placebo
Number analyzed (Participants) | 14 | 16
units on a scale (0.0 to 20.0) | 4.52 (2.81) | 6.06 (2.82)
Statistical Analysis 1: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: There is a significant difference in mean redness (i.e., mean a* number value) between the curcumin and placebo groups; Test type: Superiority or Other; p = 0.145, ANOVA

4. Secondary Outcome: Pain at Radiation Treatment Site
Description: The McGill Pain Questionnaire-Short Form (MPQ-SF) was used to determine the participants pain at treatment site. The MPQ-SF contains three subscales: affective pain, sensory pain, and perceived pain. This outcome measure compared the total pain score (range 0 to 50)and subscale scores (sensory subscale range 0 to 33; affective subscale range 0 to 12; perceived pain subscale 0 to 5) at the end of radiation therapy between the two treatment arms.
Time Frame: 4-7 weeks (prescribed course of radiation)
Population: All 30 participants that fully completed the trial were used in these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin C3 Complex | Placebo
Number analyzed (Participants) | 14 | 16
units on a scale
  MPQ Total Score | 5.71 (4.27) | 3.50 (3.43)
  Sensory Pain Subscale | 4.07 (3.29) | 2.25 (2.32)
  Affective Pain Subscale | 0.50 (0.76) | 0.50 (0.82)
  Perceived Pain Intensity | 1.14 (0.77) | 0.88 (0.62)
Statistical Analysis 1: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: There is a significant difference in mean MPQ pain scores between the curcumin and placebo groups; Test type: Superiority or Other; p = 0.218, ANCOVA; Mean Difference (Final Values) = 1.685, 95% CI 2-sided [-1.059 to 4.428]
Statistical Analysis 2: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: There is a significant difference in mean sensory subscale pain scores between curcumin and placebo groups; Test type: Superiority or Other; p = 0.152, ANCOVA; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-0.6 to 3.6]
Statistical Analysis 3: Comparison: Curcumin C3 Complex vs Placebo; Hypohesis: There is a signifcant difference in affective subscale pain scores between curcumin and placebo groups; Test type: Superiority or Other; p = 0.700, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1.1]
Statistical Analysis 4: Comparison: Curcumin C3 Complex vs Placebo; Hypothesis: There is a significant difference in mean perceived pain scores between curcumin and placebo groups; Test type: Superiority or Other; p = 0.559, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.7]

ADVERSE EVENTS:
Time Frame: The last assessment for every participant was 6 month after completion of radiation therapy. Symptom Inventory was used to monitor side effects during radiation therapy as well as in follow-up assessments. No adverse events occurred during this study.
Arm/Group | Curcumin C3 Complex | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

LIMITATIONS AND CAVEATS:
The primary limitation of this clinical study is the small sample size. This study was a pilot trial to generate an effect and sample size for a larger confirmatory trial. We accrued patients to this study until we had 30 fully evaluable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No